CLINICAL TRIAL: NCT02484872
Title: L'Inflammation A-t-elle Une Implication Significative Dans l'évolution du Cancer Bronchique?
Brief Title: Has Inflammation a Significant Implication in Lung Cancer Evolution?
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: European Lung Cancer Working Party (Other)
Collaborators: Jules Bordet Institute (Other)
Responsible Party: Sponsor
Other Study IDs: ELCWP01501
Record Dates: First submitted 2015-06-24; First posted 2015-06-30 (Estimated); Last update posted 2021-08-23 (Actual); Status verified 2021-08

CONDITIONS: Lung Neoplasms
Keywords: Inflammation; Glasgow score; Intensive Care Unit; Emergency
MeSH Terms: conditions — Lung Neoplasms; Inflammation; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood sampling (serum)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Lung neoplasms: Lung neoplasms irrespective of stage and histology

SUMMARY:
Systemic inflammation is a potential prognostic factor in cancer. Inflammation scores as the Glasgow score have been tested in cancer and specifically in lung cancer patients. The aim of the study is to look at the prognostic and predictive value of inflammation during cancer evolution, on the risk of complications leading to ICU admission and the risk of death.

DETAILED DESCRIPTION:
Patients with newly diagnosed lung cancer will be eligible. All patients will have a blood sampling allowing testing inflammation and cytokine analyses at diagnosis, during work-up and in case of complication.

ELIGIBILITY:
Inclusion Criteria:

* Lung neoplasms irrespective of stage, histology

Exclusion Criteria:

* Previously treated lung neoplasms
* A history of prior malignant tumour, except non-melanoma skin cancer or in situ carcinoma of the cervix or cured malignant tumour (more than 5 year disease-free interval)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Newly diagnosed untreated lung neoplasms
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2015-05 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Survival | Measured from diagnosis until death or last date known to be alive, or at least 48 months

SECONDARY OUTCOMES:
Complications leading to emergency/ICU | From inclusion until death, or a least 48 months
  Recording any complication leading to consultation at the emergency department or admission into the intensive care unit

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Pascale Meert, MD, PhD, Study Chair — Jules Bordet Institute
Locations (1):
- Department of Intensive Care Unit and Thoracic Oncology Institut Jules Bordet, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: Undecided